CLINICAL TRIAL: NCT02789397
Title: Clinical Trial to Assess the Efficacy of Rituximab and Azathioprine in the Treatment of Granulomatous and Lymphocytic Interstitial Lung Disease (GLILD) in Adult Patients With Common Variable Immunodeficiency (CVID)
Brief Title: Treatment of Granulomatous and Lymphocytic Interstitial Lung Disease in Patients With Common Variable Immunodeficiency
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding for study.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, John M. Routes, Professor and Chief, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO26723
Record Dates: First submitted 2016-05-16; First posted 2016-06-03 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Granulomatous and Lymphocytic Interstitial Lung Disease
Keywords: Granulomatous and lymphocytic interstitial lung disease (GLIILD); common variable immunodeficiency; Rituximab; Azathioprine; primary immunodeficiency; GLIILD; CVID
MeSH Terms: conditions — Common Variable Immunodeficiency; Primary Immunodeficiency Diseases | interventions — Rituximab; resiniferatoxin; Azathioprine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (RTX) and Azathioprine (AZA) (Active Comparator): Rituximab 375 mg/m2/dose IV over 4 hours first dose, IV over 2-3 hours each subsequent dose weekly for 4 weeks at enrollment and again at months 6 and 12. Azathioprine: Starting dose of azathioprine will be 50 mg and increased in 25 mg increments to a maximum dose of 150 mg or 2 mg/k/day (whichever is lowest) as tolerated. Azathioprine will be administered by mouth daily for 18 months.
  Interventions: Drug: Rituximab (RTX) and Azathioprine (AZA)
- Placebo (Placebo Comparator): IV placebo will be administered on the same schedule as Rituximab. Oral placebo will be administered by mouth daily for 18 months.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Rituximab (RTX) and Azathioprine (AZA) — Rituximab 375 mg/m2/dose IV over 4 hours first dose, IV over 2-3 hours each subsequent dose weekly for 4 weeks at enrollment and again at months 6 and 12 for the active comparator arm Rituximab (RTX) and Azathioprine (AZA).
  Other Names: Truxima
  Arms: Rituximab (RTX) and Azathioprine (AZA)
Drug: Placebos — IV placebo will be administered on the same schedule as Rituximab and oral placebo will be administered by mouth daily for 18 months.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This phase II study will assess the effect of a treatment combination of Rituximab and azathioprine in patients with Granulomatous and Lymphocytic Interstitial Lung Disease (GLILD) compared to placebo, based on change in lung function at 18 months compared to baseline. The researchers will also assess if the drugs improved quality of life.

DETAILED DESCRIPTION:
BACKGROUND Common Variable Immunodeficiency (CVID) is one of the most clinically important primary immunodeficiencies due to its frequency, serious complications, and long-term costs of therapy. A form of lung disease known as granulomatous and lymphocytic interstitial lung disease (GLILD) occurs in 10-15% of patients with CVID. The causes of GLILD are unknown; no long-term study has defined the natural course of GLILD; and no clinical trials have been done to define the best possible treatment for this condition. As a result, currently there is no proven standard of care for the treatment of GLILD.

The best treatment for individuals with GLILD is not currently known. Some doctors believe that GLILD does not always continue to get worse and patients should only be treated unless this happens. Other doctors believe GLILD is always progressive and should be treated early to prevent more problems later.

There is compelling evidence to support that treatment using rituximab (RTX) in conjunction with azathioprine (AZA), may improve the lung function and abnormalities seen on high resolution CT (HRCT) scans of the chest.

STUDY GROUPS Patients in this study will either receive a placebo or a combination of Rituximab and azathioprine. These drugs are approved by the US Food and Drug Administration for other conditions, but not yet for this disease.

Because no one knows which of the treatments is best, patients will be "randomized" into one of the two study groups. Randomization means that you are put into a group by chance.

TREATMENT Eligible patients will be randomized to receive either 18 months of Rituximab and Azathioprine (20 patients) or placebo (20 patients). Rituximab will be administered intravenously (IV) weekly for four consecutive weeks at enrollment and months 6 and 12. IV placebo will be administered on the same schedule as Rituximab. Azathioprine or oral placebo will be administered by mouth daily for 18 months.

SUMMARY OF STUDY PROCEDURES

-Month 1, 6, 12

Patients will be required to travel to a study site weekly for four consecutive weeks at enrollment and at 6 and 12 months to receive study infusions. At each of these visits, patients will be given:

* Your study infusions
* Physical exams with vital signs
* Blood tests to check your organ function

Every six months (Enrollment, 6, 12 & 18 months) while receiving study treatment, patients will be asked to complete the following study tests:

* Lung Function testing
* High resolution CT of the chest
* Quality of Life Questionnaire, 6-min walk distance test and Karnofsky performance scale.
* Blood for research - approximately 10 teaspoons of blood will be collected

Monthly Labs Following the first month of study treatment, patients will be required to visit their local clinic/hospital for a blood draw to monitor their lab values twice monthly for the second and third months of treatment, then monthly.

Final Study Visit

The final study visit will take place at Month 24 after start of study treatment. Patients will also have the following tests done:

* Physical exams with vital signs
* Lung Function testing
* High resolution CT of the chest
* Quality of Life Questionnaire, 6-min walk distance test and Karnofsky performance scale.
* Blood for research - approximately 10 teaspoons of blood will be collected

ELIGIBILITY:
INCLUSION CRITERIA:

Age:

* Patients must be 18 years of age or older.

Diagnosis:

* Diagnosis of CVID in accordance with international criteria which includes: A) Serum immunoglobin G (IgG) at least 2 standard deviations below the age adjusted norm; B) Decreased serum immunoglobin A (IgA) and/or immunoglobin M (IgM); C) Age > 4 years.; D) Abnormal specific antibody production in response to immunization; E) Exclusion of secondary causes of hypogammaglobulinemia.
* Diagnosis of GLILD based on histopathologic abnormalities of lung tissue obtained by open lung biopsy within 12 months of enrollment and confirmed by Pathology Core.

Performance Level:

* Karnofsky Performance Status (KPS) ≥ 50%

Prior Therapy:

* Patients must have fully recovered from the acute toxic effects of all prior therapy.
* Systemic steroids need to be completed at least 60 days from the time of enrollment.

Organ Function:

* Adequate Lung Function defined as:

  • FVC > 60 % predicted and

  • DLco > 35 % predicted
* Adequate Bone Marrow Function defined as:

  • Peripheral absolute neutrophil count (ANC) ≥ 750/mm3 and

  • Platelet count ≥ 50,000/mm3
* Adequate Hepatic Function as evidenced by:

  * Direct Bilirubin < 1.5 x upper limit of normal (ULN) for age
  * Serum glutamic pyruvic transaminase (SGPT) (ALT) < 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
* Adequate Renal Function as defined by a normal serum creatinine

Reproductive Function:

o Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.

* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of childbearing potential must agree to use an effective method of contraception approved by the investigator during the study.
* Sexually active females of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device (UD), surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 6 months after the last dose of study therapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 6 months after the last dose of study therapy.

Regulatory Requirements

* All patients must sign a written informed consent.
* All institutional, FDA, and NIH requirements for human studies must be met.

EXCLUSION CRITERIA:

Infection:

* Patients with uncontrolled infection are not eligible.
* Patients with documented serious infection within 3 months of screening or opportunistic infection within 6 months of screening are not eligible.

Cardiac Function:

o Patients cannot be diagnosed with New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias, or uncontrolled hypertension.

Allergies:

o Known hypersensitivity to any of the components of RTX or AZA.

Current Therapy:

* Systemic immunosuppressive medications including steroids.
* Steroids can be used to prevent or to treat infusion-related RTX symptoms, but this should be used only prior to or immediately after the RTX infusion, and should not be continued beyond 3 days. The use of systemic steroids should be recorded.
* Inhaled steroids are acceptable.

Previous Therapy:

o Previous treatment with RTX or AZA for GLILD.

Pregnant Females:

o Pregnant females will not be allowed to participate in this study.

Hepatic Disease:

o Known cirrhosis and/or portal hypertension.

Hepatitis B or Hepatitis C Infection:

* All patients will be screened for Hepatitis B and C by polymerase chain reaction (PCR).
* Hepatitis C positive as determined by PCR.
* Hepatitis B Reactivation: Hepatitis B Reactivation is defined as Hepatitis B carrier patients with one of the following:

  * Positive hepatitis B e-antigen (HBe-Ag)
  * Quantitative hepatitis B Viral (HBV) DNA Load > 10^5 genomes/ml

Human Immunodeficiency Virus (HIV) 1 Positive:

o HIV 1 infection will be determined by PCR.

Homozygous Mutations:

o Patients with homozygous mutations of thiopurine methyltransferase (TPMT) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
The effect of treatment with RTX/AZA in patients with GLILD compared to placebo, based on change in forced vital capacity (FVC) at 18 months compared to baseline. | Baseline and 18 months
  Pulmonary Function Tests (PFTs) will be performed to measure lung volumes and airflow for evidence of restrictive and obstructive lung disease. PFTs are used to measure lung volumes and airflow for evidence of restrictive and obstructive lung disease. Measurements will be obtained by standard techniques following guidelines outlined by the American Thoracic Society. Spirometry, during screening, needs to be done pre- and post-bronchodilator. All subsequent spirometry is done post-bronchodilator. Diffusion capacity for carbon monoxide is always done post-bronchodilator. Spirometry will be performed to access the forced expiratory volume (FEV1) and forced vital capacity (FVC). Carbon monoxide diffusion capacity will be performed to assess gas exchange.

SECONDARY OUTCOMES:
The effect of treatment with RTX/AZA relative to placebo on the changes over time in high-resolution CT scans of the chest. | Baseline, six months, 12 months, 18 months, 24 months
  Non-contrast, low dose HRCT scans of the chest will be performed at the intervals and analyzed. Studies will be performed on high-end scanners (64 or above detector rows) capable of producing thin section (1-1.25mm) lung algorithm scans.
Correlate changes in pulmonary function (FVC, FEV1, DLco) with extent of pulmonary fibrosis obtained on open lung biopsy. | 24 months
  Pulmonary Function Tests (PFTs) will measure forced vital capacity, forced expiratory volume in one second, diffusing capacity of the lungs for carbon monoxide (DLCO) (e.g., DLco will be measured by the single-breath technique using a 10-second breath hold). Histopathologic abnormalities of lung tissue will be determined by open lung biopsy.
Correlate changes in pulmonary function (FVC, FEV1, DLco) with high-resolution CT scan scores over time in the two randomized groups of patients. | 24 months
  Pulmonary Function Tests (PFTs) will measure forced vital capacity, forced expiratory volume in one second, diffusing capacity of the lungs for carbon monoxide (DLCO) (e.g., DLco will be measured by the single-breath technique using a 10-second breath hold). These will be compared with high-resolution CT scan scores.
Changes in FVC and HRCT of the chest (maintained for 6 months after completion of therapy in both randomized groups) | Baseline, six months, 12 months, 18 months and 24 months
  Pulmonary Function Tests (PFTs) will measure forced vital capacity, forced expiratory volume in one second, diffusing capacity of the lungs for carbon monoxide (DLCO) (e.g., DLco will be measured by the single-breath technique using a 10-second breath hold). High-resolution CT scans will be performed.
Incidence of lymphoma in patients treated with RTX/AZA or placebo over the time of enrollment in the study. | 24 months
  Patients will be monitored with physical examinations, laboratory tests (CBC, auto diff, ALT, bilirubin, serum creatinine, platelets, comprehensive lymphocyte phenotype and cell sort).
Changes in quality of life in the two randomized groups of patients as measured by SGRQ total score. | Baseline, six months, 12 months, 18 months and 24 months
  Quality of life will be measured by the St. George's Respiratory Questionnaire (SGRQ), a pulmonary disease specific questionnaire measuring self-reported dyspnea symptoms and their relationship to activities of daily living and psychological functioning.
Changes in quality of life in the two randomized groups of patients as measured by Karnofsky Performance Status Scale (KPS). | Baseline, six months, 12 months, 18 months and 24 months
  Karnofsky Performance Status Scale (KPS) will be performed at baseline, six months, 12 months, 18 months and 24 months.
Changes in quality of life in the two randomized groups of patients as measured by 6-minute Walking Test. | Baseline, six months, 12 months, 18 months and 24 months
  The 6-minute Walking Test will performed at baseline, six months, 12 months, 18 months and 24 months.
Dysregulated molecular pathway determined by performing whole transcriptome sequencing. | 24 Months
  This will be done by performing whole transcriptome sequencing on GLILD, idiopathic pulmonary fibrosis (IPD), sarcoidosis and normal lung tissue.
Lung transcriptome predicts response to RTX/AZA therapy (performing whole transcriptome sequencing on GLILD, IPD, sarcoidosis and normal lung tissue) and confirm that lung transcriptome predicts response to RTX/AZA therapy. | 24 Months
  This will be done by performing whole transcriptome sequencing on GLILD, IPD, sarcoidosis and normal lung tissue.
Peripheral blood biomarkers as indicators of GLILD disease activity. | 24 Months
  The research team will examine blood specimens and evaluate Human Leukocyte Antigen - DR isotype (HLA-DR) negative and positive T cells.
Presence of bacterial (16S rRNA), fungal (Internal Transcribed Spacer region/ITS) and viral sequences (unbiased high-throughput sequencing) in the lungs of GLILD patients. | 24 Months
  This will be done by screening lung biopsies from patients with GLILD, idiopathic pulmonary fibrosis, pulmonary sarcoidosis, or no known pulmonary disease.
Prevalence and abundance of bacterial, fungal and viral sequences. | 24 Months
  This will be measured with quantitative PCR analysis of lung tissues obtained from patients with GLILD, idiopathic pulmonary fibrosis, pulmonary sarcoidosis or no known lung disease.

CONTACTS AND LOCATIONS:
Overall Officials: John M Routes, MD, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zdziarski P, Gamian A. Lymphoid Interstitial Pneumonia in Common Variable Immune Deficiency - Case Report With Disease Monitoring in Various Therapeutic Options: Pleiotropic Effects of Rituximab Regimens. Front Pharmacol. 2019 Jan 18;9:1559. doi: 10.3389/fphar.2018.01559. eCollection 2018. PMID 30713498